CLINICAL TRIAL: NCT04042441
Title: A Multi-centre Prospective Non-interventional Study Investigating the Clinical Effectiveness of Ryzodeg® (Insulin Degludec/Insulin Aspart) in Patients With Type 2 Diabetes Mellitus in a Real-world Setting
Brief Title: A Research Study, Looking at How Ryzodeg® (Insulin Degludec/Insulin Aspart) Works in People With Type 2 Diabetes in Local Clinical Practice
Acronym: ARISE
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN5401-4525; U1111-1227-8654 (Other: World Health Organization (WHO))
Record Dates: First submitted 2019-07-31; First posted 2019-08-02 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin degludec, insulin aspart drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ryzodeg® as per local practice: Real-world population of patients with Diabetes Mellitus, Type 2 (T2DM), who have been initiated or switched to Ryzodeg® from previous antihyperglycaemic treatment according to local clinical practice.
  Interventions: Drug: Insulin Degludec/Insulin Aspart

INTERVENTIONS:
Drug: Insulin Degludec/Insulin Aspart — Insulin Degludec/Insulin Aspart (Ryzodeg®) as prescribed by the patient's treating physician. The decision to initiate or switch into treatment with commercially available Ryzodeg® has been made before, and independently from, the decision to include the patient in this study.

SUMMARY:
The purpose of the study is to collect information on how Ryzodeg® works in real world patients and to see if Ryzodeg® can lower blood sugar levels. Participants will get Ryzodeg® as prescribed to them by their doctor. The study will last for about 6 to 9 months. Participants will be asked questions about their health and their diabetes treatment as part of their normal doctor's appointment.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any study-related activities. Study-related activities are any procedures related to recording of data according to the protocol.
* The decision to initiate or switch into treatment with commercially available Ryzodeg® has been made by the patient/Legally Acceptable Representative (LAR) and the treating physician based on local label before, and independently from, the decision to include the patient in this study.
* Male or female, age above or equal to 18 years at the time of signing informed consent.
* Diagnosed with T2DM and treated with any anti-hyperglycaemic medication(s) other than Ryzodeg® for at least 26 weeks prior to signing informed consent.
* Available and documented HbA1c value for 12 weeks or less prior to signing informed consent.

Exclusion Criteria:

* Hypersensitivity to the active substance or to any of the excipients as specified in the Ryzodeg® local label.
* Previous participation in this study. Participation is defined as signed informed consent.
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.
* Previous treatment with Ryzodeg®.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Real-world population of type 2 patients, who have been initiated or switched to Ryzodeg® from previous antihyperglycaemic treatment according to local clinical practice
Sampling Method: Non-Probability Sample
Enrollment: 1122 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2020-12-11 (Actual); Study Completion 2020-12-11 (Actual)

PRIMARY OUTCOMES:
Change in local laboratory measured glycosylated haemoglobin (HbA1c) | From baseline (week 0) to end of study (week 26-36)
  Percentage point

SECONDARY OUTCOMES:
HbA1c less than 7% (Yes/No) | At the end of study (week 26-36)
  Percentage of patients
HbA1c less than pre-defined individual treatment target (Yes/No) | At the end of study (week 26-36)
  Percentage of patients
Change in local laboratory measured fasting plasma glucose (FPG) | From baseline (week 0) to end of study (week 26-36)
  mg/dL
Change in local laboratory measured FPG | From baseline (week 0) to end of study (week 26-36)
  mmol/L
Change in insulin dose (total, basal, prandial) | From baseline (week 0) to end of study (week 26-36)
  units/day
Change in body weight | From baseline (week 0) to end of study (week 26-36)
  Kg
Number of patient recollection of non-severe hypoglycaemic episodes | At baseline (week 0). Episodes occurring within 4 weeks prior to initiation of treatment with Ryzodeg®
  Number of episodes
Number of patient recollection of non-severe hypoglycaemic episodes | At the end of study (week 26-36). Episodes occurring within 4 weeks prior to end of study
  Number of episodes
Number of patient recollection of nocturnal non-severe hypoglycaemic episodes | At baseline (week 0). Episodes occurring within 4 weeks prior to initiation of treatment with Ryzodeg®
  Number of episodes
Number of patient recollection of nocturnal non-severe hypoglycaemic episodes | At end of study (week 26-36). Episodes occurring within 4 weeks prior to end of study
  Number of episodes
Number of patient recollection of overall severe hypoglycaemic episodes | At baseline (week 0). Episodes occurring within 26 weeks prior to initiation of treatment with Ryzodeg®
  Number of episodes
Number of patient recollection of overall severe hypoglycaemic episodes | At the end of study (week 26-36). Episodes occurring within 26 weeks prior to end of study
  Number of episodes
Number of weekly self-measured plasma glucose (SMPG) measurements | At baseline (week 0). Measurements occurring within 7 days prior to initiation of treatment with Ryzodeg®
  Number of measurements
Number of weekly self-measured plasma glucose (SMPG) measurements | At end of study (week 26-36). Measurements occurring within 7 days prior to end of study
  Number of measurements
Reason for initiating Ryzodeg® (pre-specified response option(s)) | At baseline (week 0)
  Percentage of patients per response option
Discontinue treatment with Ryzodeg® during the treatment period (Yes/No) | At treatment discontinuation (week 0-36) or at end of study (week 26-36). After initiation of treatment with Ryzodeg® until treatment discontinuation
  Percentage of patients
Reason for discontinuing treatment with Ryzodeg® during the treatment period, if applicable, (pre-specified response option(s)) | At treatment discontinuation (week 0-36). After initiation of treatment with Ryzodeg® until treatment discontinuation
  Percentage of patients per response option
Time period from initiation to discontinuation of treatment with Ryzodeg® | At treatment discontinuation (week 0-36). After initiation of treatment with Ryzodeg® until treatment discontinuation
  Days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (64):
- Australia (10):
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Illawarra Diabetes Service Clinical Trials & Research Unit, Wollongong, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Mater Hospital Brisbane, South Brisbane, Queensland
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - South Australian Endocrine Research, Keswick, South Australia
  - Hobart Cardiology, Hobart, Tasmania
  - Box Hill Specialist Consulting rooms, Box Hill, Victoria
  - Baker IDI Heart and Diabetes Institute, Melbourne, Victoria
  - Rockingham General Hospital, Cooloongup, Western Australia
- India (10):
  - Excelcare Hospital, Guwahati, Assam
  - Columbia Asia Hospital, Bangalore, Karnataka
  - Pace Diabetes Center, Bangalore, Karnataka
  - DEW Medicare & Trinity hospital, Nagpur, Maharashtra
  - Max Super Speciality Shalimar Bhagh, Delhi, New Delhi
  - AMRI Hospital, Bhubaneswar, Odisha
  - Fortis Heart Institute and Multispeciality Hospital, Mohali, Punjab
  - R.M. Diabetes Education & Research Foundation, Chennai, Tamil Nadu
  - Narayana Superspeciality Hospital, Howrah, West Bengal
  - Fortis Hospital, New Delhi
- Malaysia (14):
  - Island Hospital, George Town
  - Remedic Clinic, Kangar
  - Pantai Hospital, Kedah
  - Kota Bahru Medical Centre Sdn Bhd, Kelantan
  - Hospital Universiti Sains Malaysia, Kota Bharu, Kelantan
  - Gleneagles Hospital, Kuala Lumpur
  - Subang Jaya Medical Center, Kuala Selangor
  - Thomson Hospital, Kuala Selangor
  - Borneo Medical Centre, Kuching
  - KPJ Kuching, Kuching
  - Mahkota Medical Center, Malacca
  - Pantai Hospital Ayer Keroh, Malacca
  - Klinik Chong, Perak
  - Hospital Putrajaya, Putrajaya
- Philippines (11):
  - Panay Healthcare Medical Center, Aklan
  - Perpetual Succor Hospital, Cebu City
  - Davao Doctors Hospital, Davao City
  - Iloilo Diabetes Care Center, Iloilo City
  - Makati Medical Center, Makati City
  - University of Santo Tomas, Manila
  - Manila Doctor's Hospital, Manila
  - University of Sto. Tomas Hospital, Manila
  - St. Luke's Medical Center, Quezon City
  - Providence Hospital, Quezon City
  - University of the East-Ramon Magsaysay Memorial Medical Ctr, Quezon City
- Saudi Arabia (10):
  - King Abdulaziz University Hospital, Jeddah
  - Dr Bakhsh Hospital, Jeddah
  - Dr. Ghassan N. Faroun Hospital, Jeddah
  - Saudi German Hospital, Jeddah
  - My clinic, Jeddah
  - Umm Alquara University Hospital, Mecca
  - Specialized medical center, Riyadh
  - Riyadh Care Hospital, Riyadh
  - National Guard Hospital, Riyadh
  - Dallah Hospital, Riyadh
- South Africa (9):
  - Greenacres Hospital, Port Elizabeth, Eastern Cape
  - Netcare Greenacres Hospital, Port Elizabeth, Eastern Cape
  - ProHealth Wellness Centre, Port Elizabeth, Eastern Cape
  - Hemant Makan, Johannesburg, Gauteng
  - Dr Moosa's Rooms, Lenasia, Gauteng
  - Prof P. Joshi, Pretoria, Gauteng
  - Dr H Bacus, Berea, KwaZulu-Natal
  - Union Hospital, Alberton
  - Medi-Clinic Bloemfontein, Bloemfontein

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Result] Fulcher GR, Cohen ND, Davies K, d'Emden M, Glastras SJ, Mah PM, McCallum RW, Moses R, Thong KY, Roberts A. Initiating or switching to insulin degludec/insulin aspart in a real-world population of adults with type 2 diabetes in Australia: results from a prospective, non-interventional study. Intern Med J. 2024 Oct;54(10):1626-1633. doi: 10.1111/imj.16492. Epub 2024 Aug 22. PMID 39171857
- [Derived] Baruah MP, Aneja P, Pitale S, Bhograj A, Agrawala RK, Aggarwal A, Mahadev PG, Madhavdas DC, Shah S, John M, Pathan MKA, Revanna M, Chandrappa M, Singh KP. Initiation or switch to insulin degludec/insulin aspart in adults with type 2 diabetes in India: Results from a prospective, non-interventional, real-world study. J Family Med Prim Care. 2024 Sep;13(9):3590-3597. doi: 10.4103/jfmpc.jfmpc_1401_23. Epub 2024 Sep 11. PMID 39464932
- [Derived] Fulcher GR, Akhtar S, Al-Jaser SJ, Medina J, Mohamed M, Nicodemus NA Jr, Olsen AH, Singh KP, Kok A. Initiating or Switching to Insulin Degludec/Insulin Aspart in Adults with Type 2 Diabetes: A Real-World, Prospective, Non-interventional Study Across Six Countries. Adv Ther. 2022 Aug;39(8):3735-3748. doi: 10.1007/s12325-022-02212-3. Epub 2022 Jun 25. PMID 35752730
- [Derived] Fulcher GR, Jarlov H, Piltoft JS, Singh KP, Liu L, Mohamed M, Nicodemus NA Jr, Al-Jaser SJ, Kok A. ARISE-a prospective, non-interventional, single-arm study assessing clinical parameters associated with the use of insulin degludec/insulin aspart in patients with type 2 diabetes in real-world settings: rationale and design. Endocrine. 2021 Dec;74(3):530-537. doi: 10.1007/s12020-021-02887-8. Epub 2021 Oct 12. PMID 34637072